CLINICAL TRIAL: NCT02030873
Title: The Effect of Virtual Simulation Training With the Visible Ear Simulator on Mastoidectomy Performance of Otorhinolaryngology Trainees
Brief Title: The Effect of Virtual Simulation Training in Mastoidectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Steven Andersen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: H-4-2014-FSP-2
Record Dates: First submitted 2014-01-02; First posted 2014-01-09 (Estimated); Last update posted 2015-05-05 (Estimated); Status verified 2015-05

CONDITIONS: Medical Education; User-Computer Interface; Clinical Skills; Motor Skills; Temporal Bone
Keywords: virtual simulation; temporal bone; surgical training; medical education; self-directed learning; final product assessment; cognitive load; reaction time; skills training; simulator metrics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Virtual simulation training first (Experimental): Participants in this arm receive virtual simulation training before dissection training.
  Interventions: Other: Virtual simulation training
- Dissection training first (No Intervention): Participants in this arm receive dissection training first and then virtual simulation training.

INTERVENTIONS:
Other: Virtual simulation training — Virtual simulation training in the Visible Ear Simulator.
  Arms: Virtual simulation training first

SUMMARY:
The purpose of this study is to investigate the effect of virtual simulation training on mastoidectomy dissection performance of otorhinolaryngology trainees, to explore performance assessment using a final-product analysis approach and to explore the role of cognitive load.

DETAILED DESCRIPTION:
Traditional dissection training in temporal bone surgery is not evidence-based yet gold standard. In the recent years the Visible Ear Simulator has been used as an introduction to mastoidectomy in the Danish temporal bone course curriculum before letting the participants move on to dissection training in order to maximize the yield from the dissection training. Instructors have the impression that participants perform better in dissection after the simulator training session has been introduced. Our pilot study suggests that participants perform better in the simulator compared to traditional dissection training. This could be due to a reduction of the cognitive load in the virtual simulator.

These observations lead to the hypothesis that virtual simulation training of mastoidectomy provides an effect that improves performance in traditional dissection training.

ELIGIBILITY:
Inclusion Criteria:

* Resident in otorhinolaryngology postgraduate year 2-5
* Informed written consent

Exclusion Criteria:

* Previous participation in formal mastoidectomy training in a virtual simulator

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Change in Final Product Assessment Score | 3 hours
  Mastoidectomy final product assessment score using a modified Welling Scale for performance assessment

SECONDARY OUTCOMES:
Change in simulator metrics | 3 hours
  Integrated simulator metrics including volume drilled (inside+outside target volumes), collisions with vital structures in simulation and time.
Change in reaction time | 3 hours
  Reaction time to a visual or auditory cue (in ms)
Simulation experience | At recruitment
  Background data from a questionnaire including questions on prior simulation training and experience
Demographics | At recruitment
  Background data from a questionnaire on participant demographics.
Computer skills | At recruitment
  Background data from a questionnaire on experience and interests in computers and IT

CONTACTS AND LOCATIONS:
Overall Officials: Steven AW Andersen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark